CLINICAL TRIAL: NCT00043797
Title: Lidorestat (IDD 676) for the Treatment of Diabetic Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Institute for Diabetes Discovery, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 676/US/2-01
Record Dates: First submitted 2002-08-13; First posted 2002-08-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-12

CONDITIONS: Diabetic Polyneuropathy
Keywords: ARI; Diabetic polyneuropathy; Diabetic complications
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Complications | interventions — lidorestat

INTERVENTIONS:
Drug: Lidorestat (IDD 676)

SUMMARY:
This clinical trial is to determine an effective dosage and to study the safety of an investigational drug -lidorestat (IDD-676)- which is intended to stop or slow the progression of diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy is one of the most important and serious complications of diabetes. It can cause pain and loss of sensation, loss of mobility and lead to chronic wounds and amputations. Studies indicate 50% or more of people who have diabetes now have or will have significant neuropathy.

Several currently marketed or investigational drugs are available to treat the painful symptoms of diabetic peripheral neuropathy, but there are no approved drugs that have been shown to prevent or slow the progression of the neuropathy itself.

The current clinical trial is an early phase II study designed to investigate the safety of the investigational drug lidorestat (IDD-676) and to determine the effect of various dose levels on important biochemical processes in the pathology of diabetic neuropathy.

Participants who enter and complete this study will, if the agent is successful, help in a very important way to bring an effective treatment from research laboratories to widespread availability for treatment. On the basis of the results of this study, large scale studies will be undertaken to support application for product registration and distribution in the U.S. and other countries throughout the world.

ELIGIBILITY:
Inclusion:

* Clinical diagnosis of Type 1 or Type II diabetes with mild to moderate diabetic peripheral neuropathy.
* Healthy status except for diabetes
* Ability to make frequent clinic visits over a 7-month period.
* Willingness and ability to understand and sign consent form.

Exclusion:

* Pregnancy or breast feeding
* Presence of uncontrolled hypertension
* History or presence of significant kidney or liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (14):
- United States (11):
  - Scottsdale Medical Specialists, Scottsdale, Arizona
  - Glendale Adventist Medical Center, Glendale, California
  - Marin Endocrinology Associates, Greenbrae, California
  - Diabetes & Endocrine Associates, La Jolla, California
  - Radiant Research, Gainesville, Florida
  - University of Miami, Dept. of Diabetes, Endocrinology & Metabolism, Miami, Florida
  - Johns Hopkins University - School of Medicine, Baltimore, Maryland
  - Brody School of Medicine, East Carolina University, Greenville, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Texas, Southwest Medical Center, Dallas, Texas
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas
- Canada (3):
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - Centre de Recherche, Laval, Quebec
  - Hospital de L'Enfant-Jesus, Québec, Quebec

REFERENCES:
- See also: Click here for more information on diabetes and diabetic neuropathy — http://www.diabetes.org